CLINICAL TRIAL: NCT01587391
Title: A Randomised, Double-blind, Placebo-controlled Trial in Healthy Volunteers to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of 2.5 mg to 160 mg of BI 163538 XX
Brief Title: Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses of BI 163538 XX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1291.1; 2011-006184-22 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (2):
- BI 163538 XX (Experimental): 1 single dose per subject as oral solution
  Interventions: Drug: BI 163538 XX
- Placebo to BI 163538 XX (Placebo Comparator): 1 single dose per subject as oral solution
  Interventions: Drug: Placebo to BI 163538 XX

INTERVENTIONS:
Drug: Placebo to BI 163538 XX — 1 single dose per subject as oral solution
  Arms: Placebo to BI 163538 XX
Drug: BI 163538 XX — 1 single dose per subject as oral solution
  Arms: BI 163538 XX

SUMMARY:
To investigate safety, tolerability, pharmacokinetics including dose proportionality, and pharmacodynamics of BI 163538 XX within a predefined dose range

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects
2. overweight or obese

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | up to 15 days postdose

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 96 hours postdose
AUC0-∞ (area under the concentration-time curve of the in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours postdose
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 96 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1291.1.1 Boehringer Ingelheim Investigational Site, Neuss, Germany